CLINICAL TRIAL: NCT04087174
Title: A Phase I, Open-label, Multi-centre Study to Assess the Safety, Tolerability, and Pharmacokinetics of Capivasertib (AZD5363) in Combination With Novel Agents in Patients With Metastatic Castration Resistant Prostate Cancer
Brief Title: A Multi-centre Study to Assess the Safety, Tolerability, and Pharmacokinetics of Capivasertib (AZD5363) in Combination With Novel Agents in Patients With Metastatic Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D3618C00002
Record Dates: First submitted 2019-07-17; First posted 2019-09-12 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Prostate Cancer
Keywords: Metastatic; Castration Resistant; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — capivasertib; enzalutamide; abiraterone

STUDY DESIGN:
Intervention Model Description: The study will include up to approximately 87 evaluable patients, divided among the 4 study parts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A1: Capivasertib + enzalutamide (Experimental): From day 1 to day 28 of this study treatment, patients will continuously enroll on a starting dose of capivasertib in combination with 160 mg enzalutamide.
  Interventions: Drug: Capivasertib; Drug: Enzalutamide
- Part A1: Capivasertib dose level 1 + enzalutamide (Experimental): On day 29 of the treatment, patients will escalate the capivasertib dose to dose level+1 along with 160 mg enzalutamide.
  Interventions: Drug: Capivasertib; Drug: Enzalutamide
- Part A1: Capivasertib dose level 2 + enzalutamide (Experimental): On day 29 of the treatment, patients will escalate the capivasertib dose to dose level+2 along with 160 mg enzalutamide.
  Interventions: Drug: Capivasertib; Drug: Enzalutamide
- Part A2: Capivasertib + abiraterone (Experimental): Patients will continuously enroll on a starting dose of capivasertib in combination with 1000 mg abiraterone.
  Interventions: Drug: Capivasertib; Drug: Abiraterone
- Part B1: Capivasertib + enzalutamide (Experimental): This optional expansion will treat patients at the recommended dose regimen of capivasertib and enzalutamide.
  Interventions: Drug: Capivasertib; Drug: Enzalutamide
- Part B2: Capivasertib + abiraterone (Experimental): This optional expansion will treat patients at the recommended dose regimen of capivasertib and abiraterone.
  Interventions: Drug: Capivasertib; Drug: Abiraterone

INTERVENTIONS:
Drug: Capivasertib — Patients will receive multiple oral dose of capivasertib.
  Other Names: AZD5363
Drug: Enzalutamide — Patients will receive 160 mg oral dose of enzalutamide.
  Arms: Part A1: Capivasertib + enzalutamide; Part A1: Capivasertib dose level 1 + enzalutamide; Part A1: Capivasertib dose level 2 + enzalutamide; Part B1: Capivasertib + enzalutamide
Drug: Abiraterone — Patients will receive 1000 mg oral dose of abiraterone.
  Arms: Part A2: Capivasertib + abiraterone; Part B2: Capivasertib + abiraterone

SUMMARY:
This is a Phase Ib, open-label, multi-centre study to determine the safety, tolerability and pharmacokinetics (PK) of capivasertib when given in combination with novel agents (enzalutamide or abiraterone) to inform the selection of capivasertib dose regimens for each combination for further clinical evaluation when given to patients with metastatic castration resistant prostate cancer (CRPC). The study design allows an exploration of different doses with intensive safety monitoring to ensure the safety of the patients.

DETAILED DESCRIPTION:
The study will be conducted on multiple centers (≤10) in USA and Spain. The study design allows an exploration of different doses with intensive safety monitoring to ensure the safety of the patients.

The two planned combination treatments during Part A of this study are:

Part A1: Capivasertib and enzalutamide Part A2: Capivasertib and abiraterone Part B will include any optional dose expansion cohorts based on Safety Review Committee (SRC) review of data from Part A of this study.

The study will include up to approximately 87 evaluable patients, divided among the 4 study parts as follows:

Part A1: Up to approximately 36 patients (up to four dose levels with up to approximately 9 patients per dose level).

Part B1: Up to approximately 12 patients. Part A2: Up to approximately 27 patients (up to three dose levels with up to approximately 9 patients per dose level). Part B2: Up to approximately 12 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol prior to any mandatory study-specific procedures, sampling, and analyses.
2. Males aged 18 years and older at the time of signing the ICF.
3. Patients with documented evidence of metastatic CRPC who have had at least one line of systemic therapy for metastatic CRPC (either chemotherapy or an novel hormonal agents [NHA]) or for whom no alternative approved therapy is available.
4. World Health Organization (WHO) performance status 0 to 2 with no deterioration over the previous 2 weeks and minimum life expectancy of 12 weeks, as assessed at day 1.
5. Patients must be able to swallow and retain oral medication.
6. Agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm.

   * Sterilisation (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate).
   * Patients should use barrier contraception (ie, condoms) from the time of screening until 16 weeks after discontinuation of study treatment. It is not known whether the preclinical changes seen in the male animal reproductive organs, after treatment with capivasertib, will be fully reversible or will permanently affect the ability to produce healthy sperm following treatment. Therefore, if patients wish to father children they should be advised to arrange for collection of sperm samples prior to the start of study treatment.

Exclusion Criteria:

1. Previous enrolment in the present study.
2. Prior enzalutamide therapy in the last 8 weeks.
3. Treatment with any of the following:

   * Nitrosourea or mitomycin C within 6 weeks of the first dose of study treatment.
   * Any investigational agents or study drugs from a previous clinical study within 30 days of the first dose of study treatment.
   * Any other chemotherapy, immunotherapy, immunosuppressant medication (other than corticosteroids) or anti-cancer agents within 3 weeks of the first dose of study treatment, except hormonal therapy with luteinising hormone-releasing hormone (LHRH) analogues for medical castration in patients with prostate cancer, which are permitted.
   * Potent inhibitors or inducers or substrates of CYP3A4 within 2 weeks before the first dose of study treatment (3 weeks for St. John's wort) or sensitive substrates of CYP3A4, CYP2C9 and/or CYP2D6 with a narrow therapeutic window within 1 week prior to the first dose of study treatment.
4. Major surgery (excluding placement of vascular access) within 4 weeks of the first dose of study treatment.
5. Radiotherapy with a wide field of radiation within 4 weeks of the first dose of study treatment.
6. Clinically significant abnormalities of glucose metabolism as defined by any of the following:

   * Diabetes mellitus Type I or Type II requiring insulin treatment.
   * HbA1c ≥8.0% (63.9 mmol/mol).
7. Spinal cord compression or brain metastases unless asymptomatic, treated and stable and not requiring steroids for at least 4 weeks prior to start of study treatment.
8. Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease.
9. As judged by the investigator, any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension, active bleeding diatheses, or active infection including hepatitis B, hepatitis C, and human immunodeficiency virus. Screening for chronic conditions is not required.
10. Any of the following cardiac criteria:

    * Mean resting corrected QT interval (QTc) >470 milliseconds obtained from 3 consecutive ECGs.
    * Any clinically important abnormalities in rhythm, conduction, or morphology of a resting ECG (eg, complete left bundle branch block, 3rd degree heart block).
    * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, potential for torsades de pointes, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years-of-age, or any concomitant medication known to prolong the QT interval.
    * Clinically significant heart disease as evidenced by myocardial infarction or arterial thrombotic events in the past 6 months, severe or unstable angina, or New York Heart Association NYHA Class II to IV heart failure or cardiac ejection fraction measurement of <50%.
    * Experience of any of the following procedures or conditions in the preceding 6 months: coronary artery bypass graft, angioplasty, vascular stent, myocardial infarction, angina pectoris, congestive heart failure NYHA ≥2.
    * Uncontrolled hypotension defined as - systolic BP <90 mmHg and/or diastolic BP<50 mmHg.
    * Uncontrolled hypertension defined as - systolic BP >160 mmHg and/or diastolic BP ≥95 mmHg.
    * Cardiac ejection fraction outside institutional range of normal or <50% (whichever is higher) as measured by echocardiogram (or multi gated acquisition scan (MUGA), if an echocardiogram cannot be performed or is inconclusive).
11. With the exception of alopecia, any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Event (CTCAE) grade 1 at the time of starting study treatment.
12. Absolute neutrophil count <1.5×10^9/L.
13. Platelets <100×10^9/L.
14. Haemoglobin <9 g/dL (<5.59 mmol/L). (Note: any blood transfusion must have been >14 days prior to the determination of a haemoglobin ≥9 g/dL [≥5.59 mmol/L]).
15. Aspartate aminotransferase (AST) >2.5 times the ULN if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases. Total bilirubin >1.5 times ULN (*patients with confirmed Gilbert's syndrome may be included in the study). Elevated alkaline phosphatase (ALP) is not exclusionary if due to the presence of bone metastasis and liver function is otherwise considered adequate in the investigator's judgement.
16. Creatinine >1.5 times ULN concurrent with creatinine clearance <50 mL/min (measured or calculated by Cockcroft and Gault equation); confirmation of creatinine clearance is only required when creatinine is >1.5 times ULN.
17. Refractory nausea and vomiting, malabsorption syndrome, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of capivasertib.
18. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug, may affect the interpretation of the results, render the patient at high risk from treatment complications or interferes with obtaining informed consent.
19. History of hypersensitivity to active or inactive excipients of capivasertib or drugs with a similar chemical structure or class to capivasertib.
20. Judgement by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.
21. Evidence of dementia, altered mental status or any psychiatric condition that would prohibit understanding or rendering of informed consent.
22. Previous allogeneic bone marrow transplant or solid organ transplant.
23. Known immunodeficiency syndrome.
24. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
25. Abiraterone-specific exclusion criteria: Any restriction or contraindication based on the currently applicable approved abiraterone label that would prohibit the use of abiraterone.
26. Enzalutamide-specific exclusion criteria: Any restriction or contraindication based on the currently applicable approved enzalutamide label that would prohibit the use of enzalutamide.

Ages: 18 Years to 130 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 27 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2021-06-22 (Actual)

PRIMARY OUTCOMES:
Number of patients with dose limiting toxicity (DLT) for Part A1 | Day 1 to day 56 for Part A1
  A DLT is defined as an AE that occurs from the first dose of study treatment up to and including the last day of the DLT period (day 1 to day 56 for Part A1) that is assessed as unrelated to the disease, intercurrent illness, or concomitant medications and that, despite optimal therapeutic interventions, meets any of the criteria defined in the protocol.
Number of patients with DLT for Part A2 | Day 1 to day 28 for Part A2
  A DLT is defined as an AE that occurs from the first dose of study treatment up to and including the last day of the DLT period (day 1 to day 28 for Part A2) that is assessed as unrelated to the disease, intercurrent illness, or concomitant medications and that, despite optimal therapeutic interventions, meets any of the criteria defined in the protocol.
Number of patients with adverse events | For each treatment combination, from screening (Day -28 to -1) either for up to 1.5 years or up to 30 days follow-up period after discontinuation
  To investigate the safety and tolerability of capivasertib when given in combination with novel agents (enzalutamide and abiraterone) to patients with metastatic CRPC.

SECONDARY OUTCOMES:
Area under curve (AUC) for capivasertib to characterize pharmacokinetics (PK) for each treatment combination | For capivasertib and enzalutamide combination, full sampling on day 25 and on day 53; for capivasertib and abiraterone combination, full sampling on day 25.
  To characterise the PK of capivasertib when given in combination with novel agents.
Maximum plasma concentration (Cmax) for capivasertib to characterize PK for each treatment combination | For capivasertib and enzalutamide combination, full sampling on day 25 and on day 53; for capivasertib and abiraterone combination, full sampling on day 25.
  To characterise the PK of capivasertib when given in combination with novel agents.
Soft tissue objective response rate (ORR) and radiological ORR for efficacy analyses of capivasertib for each treatment combination | From screening (-28 Day) to every 8 weeks after cycle 1 day 1 for the first 24 weeks and every 12 weeks thereafter up to 1.5 years for each treatment combination
  To determine the preliminary signs of activity of capivasertib in combination with novel agents in this patient population.
Duration of response (DoR) for efficacy analyses of capivasertib for each treatment combination | From screening (-28 Day) to every 8 weeks after cycle 1 day 1 for the first 24 weeks and every 12 weeks thereafter up to 1.5 years for each treatment combination
  To determine the preliminary signs of activity of capivasertib in combination with novel agents in this patient population.
Percentage change in tumour size for efficacy analyses of capivasertib for each treatment combination | From screening (-28 Day) to every 8 weeks after cycle 1 day 1 for the first 24 weeks and every 12 weeks thereafter up to 1.5 years for each treatment combination
  To determine the preliminary signs of activity of capivasertib in combination with novel agents in this patient population.
Radiographic progression free survival (rPFS) for efficacy analyses of capivasertib for each treatment combination | From screening (-28 Day) to every 8 weeks after cycle 1 day 1 for the first 24 weeks and every 12 weeks thereafter up to 1.5 years for each treatment combination
  To determine the preliminary signs of activity of capivasertib in combination with novel agents in this patient population.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (5):
  - Research Site, Indianapolis, Indiana
  - Research Site, Omaha, Nebraska
  - Research Site, White Plains, New York
  - Research Site, Gettysburg, Pennsylvania
  - Research Site, Myrtle Beach, South Carolina
- Research Site, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Shore N, Mellado B, Shah S, Hauke R, Costin D, Adra N, Cullberg M, Teruel CF, Morris T. A Phase I Study of Capivasertib in Combination With Abiraterone Acetate in Patients With Metastatic Castration-Resistant Prostate Cancer. Clin Genitourin Cancer. 2023 Apr;21(2):278-285. doi: 10.1016/j.clgc.2022.11.017. Epub 2022 Nov 26. PMID 36572571
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3618C00002&attachmentIdentifier=65bd4b23-3a3b-4700-93fb-90a9f8a30575&fileName=D3618C00002_CSR_Synopsis_Redacted.pdf&versionIdentifier=
- See also: Results of this clinical trial are available on www.astrazenecaclinicaltrials.com — https://astrazenecagrouptrials.pharmacm.com/ST/Submission/View?id=25962